CLINICAL TRIAL: NCT01896661
Title: The Effect of Antihypertensive Agents Over Sleep Apnea: a Randomized Controlled Trial
Brief Title: Effect of Antihypertensive Agents Over Sleep Apnea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07572112.7.0000.5327; 12-0417 (Other: WebGPPG)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Obstructive Sleep Apnea
Keywords: Sleep apnea; Hypertension; Treatment; Diuretics; Chlorthalidone; Amlodipine
MeSH Terms: conditions — Hypertension; Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Diuretics; Chlorthalidone; Amiloride; Calcium Channel Blockers; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diuretics (Experimental): Chlorthalidone plus amiloride 25 and 5 mg daily, taking in the morning
  Interventions: Drug: Diuretics
- Calcium Channel Blockers (Active Comparator): Amlodipine 10 mg daily, taking in the morning
  Interventions: Drug: Calcium Channel Blockers

INTERVENTIONS:
Drug: Diuretics — Chlorthalidone plus amiloride 25 and 5 mg daily, taking in the morning
  Other Names: Chlorthalidone/Amiloride
  Arms: Diuretics
Drug: Calcium Channel Blockers — Amlodipine 10 mg daily, taking in the morning
  Other Names: Amlodipine
  Arms: Calcium Channel Blockers

SUMMARY:
Obstructive sleep apnea and hypertension are well-known cardiovascular risk factors. Their control could reduce the burden of heart disease across populations. There are several drugs to control hypertension, but the only consistently beneficial treatment to reduce apneas is continuous positive airway pressure. The demonstration that one drug could improve sleep apnea and hypertension would support a novel approach in the treatment of both diseases. The role of fluid retention in sleep apnea is known for several decades. The role of diuretics is well established in hypertension but was never appropriately tested in sleep apnea. Besides to test the efficacy of these drugs, this study will help to understand the mechanisms that link hypertension and sleep apnea and its treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind, clinical trial, comparing the association of Chlorthalidone plus amiloride 25 and 5 mg daily, versus amlodipine 10 mg daily as first drug option in patients older than 40 years of age with Stage I hypertension (140-159/90-99 mmHg) and moderate obstructive sleep apnea (15-30 apneas/hour of sleep). The primary outcomes will be the variation of apneas/hour and blood pressure. The secondary outcomes will be adverse events, somnolence scale (Epworth), ventilatory parameters and C reactive protein. The follow up will last 8 weeks. The sample size will be of 29 participants per group. The project was approved by the Ethics committee of our institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 40 years of age
* Stage I hypertension (140-159/90-99 mmHg) and moderate obstructive sleep apnea (10-40 apneas/hour of sleep)

Exclusion Criteria:

* Low life expectancy
* Other indications for the use of diuretics or calcium channel blocker -Intolerance or contraindications to the study drugs
* Pregnancy
* Established cardiovascular disease (myocardial infarction
* Stroke
* Heart failure)
* Use of more than one drug for hypertension
* Secondary hypertension
* Participation in other clinical trial in previous 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | 8 weeks
  Number of apneas/hour
Blood Pressure | 8 weeks

SECONDARY OUTCOMES:
Adverse events | 8 weeks
Somnolence scale (Epworth) and ventilatory parameters | 8 weeks
C reactive protein | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Flavio D Fuchs, MD, PhD, Study Chair — Hospital de Clinicas de Porto Alegre, Universidade Federal do Rio Grande do Sul; Fabio T Cichelero, MD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cichelero FT, Fuchs SC, Jorge JA, Martinez D, Oliveira GPF, Lucca MB, Oliveira ACT, Fuchs FD. Effect of antihypertensive agents on sleep apnea and ambulatory blood pressure in patients with hypertension: A randomized controlled trial. Sleep Med. 2024 Jul;119:417-423. doi: 10.1016/j.sleep.2024.05.035. Epub 2024 May 16. PMID 38781664
- [Derived] Cichelero FT, Martinez D, Fuchs SC, Gus M, Moreira LB, Fuchs FD. The effect of antihypertensive agents on sleep apnea: protocol for a randomized controlled trial. Trials. 2014 Jan 2;15:1. doi: 10.1186/1745-6215-15-1. PMID 24382030